CLINICAL TRIAL: NCT06175819
Title: Efficacy of Manuka Honey Nano-Formulatin on the Clinical Improvement and Inflammatory Markers Reduction in Patients With Acne Vulgaris
Brief Title: Efficacy of Manuka Honey Nano-Formulation in the Treatment of Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Maha khalifa, Associate Professor, Pharmaceutics Department, Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Manuka honey nanoformulation
Record Dates: First submitted 2023-11-19; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Prospective interventional randomized clinical trial
Who Masked: Participant
Masking Description: The intervention of each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manuka nanoformulation group (Experimental): This group will apply Manuka honey ( MgO 850, UMF+20) nanoformulation on the face lesions 2 times daily for 28 days or cure of lesions (Arm 1)
  Interventions: Other: Manuka honey( MgO 850, UMF+20) loaded nano-formulation
- Manuka honey gel group (Experimental): This group will apply Manuka honey ( MgO 850, UMF+20) gel on the face lesions 2 times daily for 28 days or cure of lesions (Arm 2)
  Interventions: Other: Manuka honey( MgO 850, UMF+20) loaded nano-formulation
- clindamycin commercial gel (Active Comparator): This group will apply clindamycin commercial gel (Clindamycin 1%gel,European pharmaceuticals, Alex, Egypt) on the face lesions 2 times daily for 28 days or cure of lesions (Arm 3)
  Interventions: Other: Manuka honey( MgO 850, UMF+20) loaded nano-formulation

INTERVENTIONS:
Other: Manuka honey( MgO 850, UMF+20) loaded nano-formulation — Assessment of the efficacy of manuka-loaded nano-formulation and manuka honey-loaded gel on the improvement of acne vulgaris
  Other Names: Manuka honey ( MgO 850, UMF+20)loaded gel

SUMMARY:
The present study aims to manufacture manuka honey-loaded nano-formulation using natural materials as a potent tissue-healing remedy and compare it to commercially available antimicrobial therapy in order to reduce the severity and recurrences of skin lesions.

DETAILED DESCRIPTION:
It was found that patients with acne suffer from lower self-esteem, depression, anxiety, and social isolation as a result of papules, pustules, nodules, cysts, and scarring. Moreover, a common complication of acne is residual post-inflammatory hyperpigmentation and acne scaring which cause further psychological and social distress. Collectively, these factors explain the reduction of quality of life .

The intervention for AV treatment has been unaltered throughout last years. There is a global shift from antibiotics concerning limiting their use due to increasing antibiotic resistance. Hence, it is imperative to provide natural products as another modality of treatment.

Manuka honey (MH) is a mono-floral honey harvested by honeybees (Apis mellifera) after pollinating and collecting nectar primarily from the Manuka tree. MH's anti-inflammatory and broad-spectrum antibacterial activity is due to its major ingredients, hydrogen peroxide H2O2 produced enzymatically, non-peroxidase methylglyoxal (MGO), and the peptide bee defensin-1 which has antimicrobial action. Furthermore, MH inhibits bacterial growth by high osmolality and low pH. A high MGO content MH nano-formulation will be fabricated to serve as a vehicle for its topical delivery.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate acne vulgaris patients.Patients will be assessed for severity of acne by Global acne grading system (GAGS).
* Age of patients: 18-40 years.
* Sex: both sexes.

Exclusion Criteria:

* Pregnancy and lactation.
* severe acne vulgaris.
* exogenous acne as industrial or cosmetic causes.
* Patients with photodermatitis or allergic dermatitis.
* serious or systemic illnesses such as liver and renal dysfunction.
* Patients with radiotherapy, cryotherapy, cutaneous malignant tumors, and patients suffer from mental illnesses.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-04-11 (Estimated); Study Completion 2024-09-11 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | 4 weeks
  Clinical evaluation: (Yun Chen MM et al.,2023)
  * cure :Reduction of lesion area ≥90%
  * Significant effect: The lesion area was reduced by 60%-89%
  * Effective: Skin lesion area reduced by 30%-59%
  * Invalid: Reduction of lesion area ≤29%
  * cure :Reduction of lesion area ≥90%
  * Significant effect: The lesion area was reduced by 60%-89%
  * Effective: Skin lesion area reduced by 30%-59%
  * Invalid: Reduction of lesion area ≤29%
Acne severity evaluation | 4 weeks
  Acne severity evaluation :
  The skin lesion scores were calculated before treatment and 4 weeks after treatment according to Global acne grading system (GAGS). (Yun Chen MM et al.,2023).

SECONDARY OUTCOMES:
Specific parameters (interleukin-1 beta ) (IL-1β)measurement | 4 weeks
  A venous Plasma samples will be obtained from all patients at first visit and after 4 weeks of treatment.
  The assay will be done using commercially available enzyme-linked immunosorbent assay (ELISA) kits before and after 4 weeks of treatment.
  The assay will be performed according to the manufacturer's instructions.
Specific parameter interleukin-17 (IL-17) measurement | 4 weeks
  A venous Plasma samples will be obtained from all patients at first visit and after 4 weeks of treatment.
  The assay will be done using commercially available enzyme-linked immunosorbent assay (ELISA) kits before and after 4 weeks of treatment.
  The assay will be performed according to the manufacturer's instructions
Specific parameter C-reactive protein (CRP) measurement | 4 weeks
  A venous Plasma samples will be obtained from all patients at first visit and after 4 weeks of treatment.
  The assay will be done using commercially available enzyme-linked immunosorbent assay (ELISA) kits before and after 4 weeks of treatment.
  The assay will be performed according to the manufacturer's instructions

CONTACTS AND LOCATIONS:
Overall Officials: Maha Khalifa, Study Director — Associate professor of pharmaceutics